CLINICAL TRIAL: NCT04959344
Title: Safety and Immunogenicity of a Klebsiella Pneumoniae Tetravalent Bioconjugate Vaccine (Kleb4V) Administered to Healthy Adults: A FTIH Phase I/II Randomized and Controlled Study
Brief Title: Safety and Immunogenicity of a Klebsiella Pneumoniae Tetravalent Bioconjugate Vaccine (Kleb4V)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Kleb4V01
Record Dates: First submitted 2021-06-25; First posted 2021-07-13 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Klebsiella Pneumoniae Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Kleb4V target dose (Experimental): Study participants receive 2 target doses of the non-adjuvanted investigational product 2 months apart.
  Interventions: Biological: Kleb4V target dose
- Kleb4V target dose + AS03 (Experimental): Study participants receive 2 target doses of the adjuvanted investigational product 2 months apart.
  Interventions: Biological: Kleb4V target dose + AS03
- Kleb4V low dose (Experimental): Study participants receive 2 low doses of the non-adjuvanted investigational product 2 months apart.
  Interventions: Biological: Kleb4V low dose
- Kleb4V low dose + AS03 (Experimental): Study participants receive 2 low doses of the adjuvanted investigational product 2 months apart.
  Interventions: Biological: Kleb4V low dose + AS03
- Placebo (Diluent) (Placebo Comparator): Study participants receive 2 doses of the Placebo 2 months apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Kleb4V target dose — Two doses of the non-adjuvanted Kleb4V target dose will be administered intramuscularly 2 months apart
  Arms: Kleb4V target dose
Biological: Kleb4V target dose + AS03 — Two doses of the adjuvanted Kleb4V target dose will be administered intramuscularly 2 months apart
  Arms: Kleb4V target dose + AS03
Biological: Kleb4V low dose — Two doses of the non-adjuvanted Kleb4V low dose will be administered intramuscularly 2 months apart
  Arms: Kleb4V low dose
Biological: Kleb4V low dose + AS03 — Two doses of the adjuvanted Kleb4V low dose will be administered intramuscularly 2 months apart
  Arms: Kleb4V low dose + AS03
Biological: Placebo — Two doses of the Placebo will be administered intramuscularly 2 months apart
  Arms: Placebo (Diluent)

SUMMARY:
In this study, the tetravalent bioconjugate candidate vaccine Kleb4V will be tested to obtain first-time-in-human (FTIH) data on its safety and immunogenicity in healthy adults.

DETAILED DESCRIPTION:
Kleb4V is a tetravalent bioconjugate vaccine including O antigen-polysaccharides of the most predominant Klebsiella pneumoniae serotypes, which will be formulated with or without Adjuvant System, AS03. Study participants will be randomized towards Kleb4V Low dose with or without AS03, Kleb4V Target dose with or without AS03, or placebo.

The study will be conducted in two steps. In Step1 (safety cohort): safety and tolerability of Kleb4V without and with Adjuvant AS03 will be evaluated first in adults of 18-40 y, and subsequently in the target population of older adults 55-70 y. Enrolment will be staggered in groups of small numbers to the different doses and formulations.

In Step 2 (target cohort): Older adults (55-70y) will be concomitantly randomized to receive 1 of the 4 different vaccine formulations or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health by medical history, laboratory findings and physical examination before receiving vaccination as judged by the investigator (subjects with a minor controlled illness, such as mild controlled hypertension, asthma or COPD (Chronic Obstructive Pulmonary Disease), and without fever may be enrolled at the discretion of the investigator)
2. Subject who is willing and able to comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits)
3. Signed written informed consent obtained from the subject
4. For Step 1 Groups 1 and 2 only: Female or male between 18-40 years (inclusive) of age
5. For Step 1 Groups 3 to 6, and Step 2: Female or male subjects between 55-70 (inclusive) years of age at the time of first vaccination
6. Female subjects of childbearing potential are eligible, as long as they practice adequate contraceptive measures from 2 months before the first vaccination until 1 month after the last vaccination.

Exclusion Criteria:

1. Health condition that, in the opinion of the investigator, may interfere with optimal participation in the study or place the volunteer at increased risk of adverse events (AEs) Study clinicians, in consultation with the principal investigator, will use clinical judgement on a case-by-case basis to assess safety risks under this criterion
2. Any clinically significant deviation from the normal range in biochemistry or hematology blood tests in the opinion of the investigator
3. Clinically significant abnormalities on physical examination
4. Suspected or known hypersensitivity (including allergy) to any of the vaccine components or to medicinal products or medical equipment whose use is foreseen in this study
5. History of allergy to any vaccine
6. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws (e.g. coagulation disorder)
7. Acute or chronic, clinically significant cardiovascular, pulmonary, hepatic or renal abnormality diseases and/or insufficiency as determined by physical examination or laboratory tests. In particular: unstable current or history of coronary artery disease or cardiac insufficiency, uncontrolled hypertension, clinically significant history of myocardial infarction, atrial fibrillation, uncontrolled or clinically significant type 2 diabetes, current or history of rheumatoid arthritis or temporal arteritis, current acute or chronic active pulmonary diseases.

   Note: Subjects may be on chronic or as needed medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition
8. Known or suspected impairment of immunological function, documented Human Immunodeficiency Virus (HIV) infection, asplenia/splenectomy, or history of autoimmune disease or lymphoproliferative disorder
9. Positive blood test for HBsAg, HCV (Hepatitis C Virus), HIV-1/2
10. Positive test for SARS-CoV-2 (severe acute respiratory syndrome coronavirus type 2)
11. History of systemic administration of immunosuppressive drugs, i.e. corticosteroids, (PO/IV/IM) within the last 4 weeks prior to 1st vaccination or for more than 14 consecutive days within 3 months prior to 1st vaccination, until the last blood sampling visit (i.e. prednisone or equivalent ≥20 mg/day). Inhaled and topical steroids are allowed.
12. Administration of anti-neoplastic and immune-modulating agents or chemotherapy within 90 days prior to informed consent
13. Planned administration of a vaccine not foreseen by the study protocol within 4 weeks prior to 1st vaccination and 4 weeks after last vaccination. Vaccination against seasonal influenza virus (or CoVID (Coronavirus disease) vaccine if on the market) is allowed outside of +/- 7 days from each vaccination
14. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational interventional vaccine/product (pharmaceutical product)
15. Body Mass Index (BMI) <19 and >30
16. History of any chronic or progressive disease that according to judgement of the investigator could interfere with the study outcomes or pose a threat to the participant's health
17. Received an investigational or non-registered product (medicinal drug or vaccine), other than the study vaccine within 3 months prior to 1st administration of study vaccine, or planned use during the study period
18. Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine
19. Blood donation of at least 500 mL blood draw within 3 months preceding injection or planned during the study period as reported by subject
20. Use of any antibiotic therapy within 1 week preceding each injection
21. Subjects with an elective surgical intervention, planned during the study period until 30 days after 2nd vaccination
22. Females lactating, or pregnancy or intention to become pregnant as reported by subject
23. Current and/or history of chronic alcohol consumption and/or drug abuse
24. History of immune-mediated disease (see Table of pIMDs (potential Immune Mediated Diseases) in Annex).
25. Heavy smokers (> 20 cigarettes per day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Safety: Occurrence, severity and relationship of solicited local and general AEs (Adverse Events) | during 7 days following each vaccination
  Occurrence, severity and relationship of solicited local and general AEs (Adverse Events)
Safety: Occurrence, severity and relationship of unsolicited AEs | during 28 days following each vaccination
  Occurrence, severity and relationship of unsolicited AEs
Safety: Occurrence, severity and relationship of medically relevant AEs, AESIs and SAEs | through the study completion, on average of 1 year
  Occurrence, severity and relationship of medically relevant AEs, AESIs (Adverse Events of Special Interest) and SAEs (Serious Adverse Events)
Immunogenicity: IgG (Immunoglobulin G) titers against the Klebsiella pneumoniae O serotypes included in the vaccine | between baseline and 28 days after the second injection
  For each active group vs. placebo: Comparison of geometric mean titers (GMTs) of serum IgG against the four K. pneumoniae O-serotypes included in Kleb4V.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Alaimo, Study Director — LimmaTech Biologics AG; Steffen Haffner, Dr, Principal Investigator — Nuvisan GmbH
Locations (2):
- Germany (2):
  - Nuvisan GmbH, Standort Gauting, Robert-Koch-Allee 29, Gauting
  - Nuvisan GmbH, Standort Neu-Ulm, Wegenerstrasse 13, Neu-Ulm

REFERENCES:
- [Derived] Alaimo C, Karaky N, Lawrence R, Bownes E, Haffner S, Kowarik M, Goldblatt D, Martin P. Safety and immunogenicity of a Klebsiella pneumoniae tetravalent bioconjugate vaccine (Kleb4V) administered to healthy adults: A first time in human phase I/II randomised and controlled study. J Infect Dis. 2025 Nov 25:jiaf600. doi: 10.1093/infdis/jiaf600. Online ahead of print. PMID 41289032
- [Derived] Chen Z, Gou Q, Yuan Y, Zhang X, Zhao Z, Liao J, Zeng X, Jing H, Jiang S, Zhang W, Zeng H, Huang W, Zou Q, Zhang J. Vaccination with a trivalent Klebsiella pneumoniae vaccine confers protection in a murine model of pneumonia. Vaccine. 2024 Oct 3;42(23):126217. doi: 10.1016/j.vaccine.2024.126217. Epub 2024 Aug 19. PMID 39163713